CLINICAL TRIAL: NCT00287131
Title: Adoptive Cell Therapy Following Non-myeloablate Chemotherapy in Metastatic Melanoma Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-04-3518-JS-CTIL
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; metastatic melanoma; adoptive immunotherapy; IL-2
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Procedure - Adoptive cell transfer — Procedure - Adoptive cell transfer

SUMMARY:
Metastatic melanoma is an aggressive and highly malignant cancer. The five-year survival rate of patients with metastatic disease is less than 5% with a median survival of only 6-10 months. Drugs like Dacarbazin (DTIC) as a single agent or in combination with other chemotherapy agents, have a response rate of 15-30%, but the duration of response is usually short, with no impact on survival. Interleukin-2 (IL-2) based immunotherapy has shown more promising results. This form of therapy has a similar response rate with some patients achieving a durable complete response. Recently the National Institute of Health (NIH) reported that by using lympho-depleting chemotherapy, followed by an adoptive transfer of large numbers of anti-tumor specific tumor-infiltrating lymphocytes (TIL), an objective regression was achieved in 51% of patients with metastatic melanoma.

Objectives: To introduce the TIL technology to advanced metastatic melanoma patients in Israel.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Melanoma patients failing to prior chemo and immunotherapy with good performance status.

Exclusion Criteria:

* Brain mets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Response rate and toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Schachter, MD, Principal Investigator — Head, Ella Institute, Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Tel Hashomer, Israel

REFERENCES:
- [Result] Besser MJ, Shapira-Frommer R, Treves AJ, Zippel D, Itzhaki O, Hershkovitz L, Levy D, Kubi A, Hovav E, Chermoshniuk N, Shalmon B, Hardan I, Catane R, Markel G, Apter S, Ben-Nun A, Kuchuk I, Shimoni A, Nagler A, Schachter J. Clinical responses in a phase II study using adoptive transfer of short-term cultured tumor infiltration lymphocytes in metastatic melanoma patients. Clin Cancer Res. 2010 May 1;16(9):2646-55. doi: 10.1158/1078-0432.CCR-10-0041. Epub 2010 Apr 20. PMID 20406835
- [Derived] Nissani A, Lev-Ari S, Meirson T, Jacoby E, Asher N, Ben-Betzalel G, Itzhaki O, Shapira-Frommer R, Schachter J, Markel G, Besser MJ. Comparison of non-myeloablative lymphodepleting preconditioning regimens in patients undergoing adoptive T cell therapy. J Immunother Cancer. 2021 May;9(5):e001743. doi: 10.1136/jitc-2020-001743. PMID 33990415
- [Derived] Itzhaki O, Jacoby E, Nissani A, Levi M, Nagler A, Kubi A, Brezinger K, Brayer H, Zeltzer LA, Rozenbaum M, Vernitsky H, Markel G, Toren A, Avigdor A, Schachter J, Besser MJ. Head-to-head comparison of in-house produced CD19 CAR-T cell in ALL and NHL patients. J Immunother Cancer. 2020 Mar;8(1):e000148. doi: 10.1136/jitc-2019-000148. PMID 32152221
- [Derived] Nemlich Y, Greenberg E, Ortenberg R, Besser MJ, Barshack I, Jacob-Hirsch J, Jacoby E, Eyal E, Rivkin L, Prieto VG, Chakravarti N, Duncan LM, Kallenberg DM, Galun E, Bennett DC, Amariglio N, Bar-Eli M, Schachter J, Rechavi G, Markel G. MicroRNA-mediated loss of ADAR1 in metastatic melanoma promotes tumor growth. J Clin Invest. 2013 Jun;123(6):2703-18. doi: 10.1172/JCI62980. PMID 23728176